CLINICAL TRIAL: NCT04288531
Title: Observational Study on the Impact of Iodine Supplementation on Maternal and Child's Thyroid Hormone Homeostasis and on the Child's Psychomotor Development, in the Portuguese Minho Region (IodineMinho)
Brief Title: Iodine Impact on Thyroid Function and Psychomotor Development, Observational Study in the Portuguese Minho Region
Acronym: IodineMinho
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minho (Other)
Collaborators: Instituto Nacional de Saúde Dr Ricardo Jorge, Portugal (Unknown); Clinical Academic Center (2CA-Braga) (Other); Hospital de Braga (Other); Administração Regional de Saúde do Norte, Portugal (Other)
Responsible Party: Principal Investigator, Joana Almeida Palha, Professor, University of Minho
Other Study IDs: UMinho-IodineMinho; U1111-1247-2293 (Other: World Health Organization)
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Iodine Deficiency; Thyroid; Pregnancy Related; Psychomotor Impairment; Hypothyroidism in Pregnancy; Nutrient Deficiency
Keywords: Iodine; Human milk; Maternal health; Nutritional assessment; Thyroid hormones; Pregnancy; Population health; Congenital hypothyroidism; Psychomotor development
MeSH Terms: conditions — Thyroid Diseases; Psychomotor Disorders; Congenital Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, Milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Pregnant and pregnant to be on iodine supplementation: Women in preconception, pregnant and lactating, receiving iodine supplementation
  Interventions: Dietary Supplement: Iodine supplementation
- Pregnant and pregnant to be not on iodine supplementation: Women in preconception, pregnant or lactating, not receiving iodine supplementation
- Women of childbearing age: Women of childbearing age not planning to become pregnant.

INTERVENTIONS:
Dietary Supplement: Iodine supplementation — Recommendation, issued by the National Health Authorities, on supplementing with iodine (200 ug/day) women during preconception, pregnancy and lactation.
  Groups: Pregnant and pregnant to be on iodine supplementation

SUMMARY:
Full intellectual capabilities are achieved only if crucial nutrients are present during development. Iodine deficiency is the most common cause of preventable brain harm in infants. Because of its critical need during pregnancy, several countries implemented programs of iodine supplementation in preconception and pregnancy. In 2013, the prevalence of iodine deficiency in Portugal has led health authorities to issue a recommendation for iodine supplementation. This study aims to evaluate the impact of iodine supplementation on maternal and fetal iodine status and thyroid function, obstetric outcomes, quality of breast milk and child psychomotor development. It also intends to evaluate whether the time of iodine supplementation initiation influences all the above-mentioned parameters. The novelty and relevance of this study reside on the number of women/child and on the extent of health parameters that will be evaluated. The information collected will contribute to the detailed characterization of thyroid hormone homeostasis throughout pregnancy and its relationship with iodine supplementation (including time of initiation). The data will provide evidence on whether this iodine supplementation strategy impacted on iodine sufficiency of the mother and the newborns, or if it needs re-evaluation.

DETAILED DESCRIPTION:
Iodine is essential for intellectual development. Its deficiency, alone, is the most frequent cause of preventable brain harm in infants. Iodine is required to synthesize thyroid hormones, key components of central nervous system development. Because of its relevance in pregnancy, several countries have implemented iodine supplementation programs in preconception, pregnancy and lactation.

Iodine deficiency has been previously shown in women of childbearing age in Portugal. Because of this, since 2013 the National Health Authorities have recommended supplementing iodine (200 ug/day) in preconception, pregnant and lactating women. However, the latest Cochrane review on the subject does not allow to conclude on whether iodine supplementation strategies implemented to date are efficient. Therefore, this study is of great public health interest.

The objectives are to:

* Evaluate whether the new policy of recommending iodine supplementation in preconception, throughout pregnancy and during lactation impacted on the prevalence of iodine deficiency in the Minho region of Portugal when compared to the same population before the recommendation.
* Evaluate whether the time of initiation of iodine supplementation (if any) influences the serum levels of thyroid hormones in the three trimesters of pregnancy.
* Evaluate whether the serum levels of thyroid hormones in the first trimester of pregnancy predict psychomotor development of the newborn at 12 months of age.

To achieve these aims the investigators will follow: i) 304 women longitudinally, before, during the three trimesters of pregnancy (primary care Health Centres), at delivery and three months after delivery, ii) their children at birth, 3 and 12 months of age; ii) perform a detailed evaluation of parameters of thyroid function (mother and child) and of psychomotor development of the newborns.

Investigators expect to provide detailed characterization of thyroid hormone homeostasis before and throughout pregnancy, their relation with iodine supplementation (and its timing of administration, if any) and with thyroid hormone parameters and psychomotor development of the newborn.

With 6 years passed since the beginning of recommendation on iodine supplementation, this is an appropriate time to assess its effectiveness. The high number of samples and parameters to analyze make this a high-power study to support public health policies.

ELIGIBILITY:
Inclusion Criteria:

* Women of who intend to become pregnant or are pregnant, able to read, write and provide informed consent

Exclusion Criteria:

* Women transferred from outside the study health centres during pregnancy and women taking iodine supplementation before recruitment.
* Women not intending to deliver at Hospital de Braga.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women from community health centers who intend to become pregnant or become pregnant and intend to delivery in the Hospital de Braga.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of iodine deficiency in pregnant women and in women of childbearing age in the Minho region | At baseline in women recruited for pregnancy follow-up and in women in childbearing age not planning to become pregnant.
  Urinary iodine.
Impact of iodine supplementation on maternal serum parameters of thyroid function and urinary iodine in the first trimester of pregnancy | First trimester of pregnancy
  Serum thyroid hormones (TSH, total and free T4, total and free T3, thyroxine-binding globulin, human chorionic gonadotropin, thyroglobulin, anti-thyroglobulin, anti-thyroperoxidase), urinary iodine.
Bayley scale assessed psychomotor development at one year of age | One year of age
  Bayley psychomotor development scale

SECONDARY OUTCOMES:
Serum parameters of thyroid function, urinary iodine and thyroid ultrasound characterization throughout pregnancy | Serum thyroid hormones and urinary iodine before iodine supplementation (if any), 1st, 2nd, 3rd trimesters of pregnancy, after delivery. Thyroid ultrasound at baseline, 3rd trimester and 3 months after delivery.
  Serum thyroid hormones (TSH, total and free T4, total and free T3, thyroxine-binding globulin, human chorionic gonadotropin, thyroglobulin, anti-thyroglobulin, anti-peroxidase), urinary iodine, thyroid ultrasound.
Serum parameters of thyroid function, urinary iodine and thyroid ultrasound characterization of newborns | One to 3 days of age (if full term babies), 1 to 3 days and 4th week of age (in premature and low birth weight babies).
  Serum thyroid hormones (TSH and eventually total and free thyroxine as retrieved from the neonatal newborn screening) and urinary iodine.
Iodine and energy composition of human milk 3 months after delivery | Three months after delivery
  Iodine and energy composition (total proteins, lipids and carbohydrates).
Fetal heart rate and thyroid volume at age 3 months | Fetal cardiotocography at 36-40 weeks of gestation and thyroid ultrasound at 3 months of age.
  Fetal cardiotocography and thyroid ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Joana A Palha, PhD, Principal Investigator — School of Medicine, University of Minho
Locations (10):
- Portugal (10):
  - Usf Maxisaude, Braga
  - Usf Braga Norte, Braga
  - Usf Ruães, Braga
  - Usf S. Lourenço, Braga
  - Usf Gualtar, Braga
  - Usf + Carandá, Braga
  - Usf Manuel Rocha Peixoto, Braga
  - Usf Bracara Augusta, Braga
  - Usf Do Minho, Braga
  - Usf S. João de Braga, Braga

IPD SHARING:
Plan to Share IPD: Yes
Data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Data will be provided for collaborative research purposes and for health authorities for public health recommendations. The Principal Investigator, research team and institution directive board will review the requests.

REFERENCES:
- [Derived] Lopes-Pereira M, Roque S, Costa P, Quialheiro A, Santos NC, Goios A, Vilarinho L, Correia-Neves M, Palha JA. Impact of iodine supplementation during preconception, pregnancy and lactation on maternal thyroid homeostasis and offspring psychomotor development: protocol of the IodineMinho prospective study. BMC Pregnancy Childbirth. 2020 Nov 13;20(1):693. doi: 10.1186/s12884-020-03376-y. PMID 33187482